CLINICAL TRIAL: NCT06111248
Title: Evaluation of the Impact of Training Healthcare Teams (Quality Improvement Project) in the Combined Use of AoA Carestation Software and Digital Intraoperative Monitoring Tools (State Entropy, Surgical Pleth Index and Train-of-Four) During General Anesthesia for Intermediate- or Major-risk Surgery on Patient Morbidity and Mortality at 28 Days
Brief Title: Impact of Training on the Use of Software and Digital Monitoring Tools During General Anesthesia for Intermediate/Major-risk Surgery on Morbidity and Mortality at 28 Days
Acronym: AoA QUALITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CIVI/2023/PC-01
Record Dates: First submitted 2023-10-20; First posted 2023-11-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: All Conditions Requiring Non-cardiac Surgery
Keywords: Anesthesia; Monitoring; Cardiovascular assessment; Anesthesiology Devices; Diagnostic and Monitoring Devices
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Prospective interventional monocentric before-and-after clinical study to evaluate the impact of a "quality improvement project" intervention. The intervention consists in informing, training and coaching teams on how to use the surgical plethysmographic index, state entropy and train-of-four intraoperative monitors and AoA software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 638 patients receiving the usual, standard management for anesthesia when undergoing surgery lasting > 60 min and involving intermediate or major non-cardiac risk.
- Experimental group (Experimental): 638 patients undergoing surgery lasting > 60 min and involving intermediate or major non-cardiac risk who have been managed by staff trained in the use of surgical plethysmographic index (SPI) state entropy (SE) and train-of-four (TOF) intraoperative monitors and AoA software.
  Interventions: Other: Training

INTERVENTIONS:
Other: Training — Staff training on the use of surgical plethysmographic index (SPI) state entropy (SE) and train-of-four (TOF) intraoperative monitors and AoA software.
  Arms: Experimental group

SUMMARY:
Tools such as surgical plethysmographic index, state entropy, train-of-four monitors exist to optimize the conduct of general anesthesia in intermediate and major risk surgery as defined by the 2022 European Society of Cardiology Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery. Although these monitors are available on anesthesia machines they are still under-used by teams due to lack of training, practice and a real understanding of their usefulness (operation, expected benefits). When used in conjunction with General Electric's AoA Carestation Insight software, these tools could have a real impact on morbidity and mortality at 28 days post-op. The aim of this prospective monocentric interventional "before/after" study is to assess the impact of training and encouraging teams to use these tools.

DETAILED DESCRIPTION:
Recently, complex monitoring tools (nociception by surgical plethysmographic index monitoring, curare by train-of four monitoring, depth of anesthesia by state entropy monitoring) have been developed to optimize the conduct of general anesthesia in intermediate and major risk surgery (surgery defined by the 2022 European Society of Cardiology Guidelines on cardiovascular assessment and management of patients undergoing non-cardiac surgery). In practice, these monitors optimize nociception and the depth of anesthesia, "neither too strong nor too light". These monitors are currently available on our anesthesia machines and can be used routinely. However, these monitors are under-used by teams due to lack of training, practice and real understanding of their usefulness (operation, expected benefits).

Excess nociception and depth of anesthesia are correlated with more postoperative complications, but no studies have ever shown that the combined use of these monitors (surgical plethysmographic index, state entropy, train-of-four) could significantly reduce postoperative morbidity and mortality in patients by optimizing the management of general anesthesia. Software (AoA Carestation insight, General Electric) connected to these monitors can :

* automatically query the use of intraoperative monitors;
* perform usage audits to monitor teams' adherence to their practices;
* coach teams by encouraging them to perform anesthesia while maintaining surgical plethysmographic index (SPI), state entropy (SE) and train-of-four (TOF) values within the thresholds considered in the literature as being optimal for anesthesia (formalized expert recommendations from the SFAR (Société Francaise d'Anesthésie et de Réanimation).

In a prospective monocentric interventional "before/after" study, the aim is to assess the impact of training and encouraging teams to use the AoA Carestation Insight software in conjunction with SPI, SE and TOF monitoring, on morbidity and mortality at 28 days post-op.

The hypothesis is that training and encouraging teams ("quality improvement project") to use these intraoperative monitoring tools (SPI, TOF, SE) during general anesthesia for intermediate- or major-risk surgery could significantly reduce 28-day morbidity and mortality (composite criterion).

ELIGIBILITY:
Inclusion Criteria:

* Patients with an ASA score 2-4.
* Patients due to be operated on under general anesthesia for any intermediate- or major-risk non-cardiac procedure lasting > 60 min.
* Patients affiliated to, or benefiting from, a health insurance plan.

Exclusion Criteria:

* Patients who have indicated their refusal to participate in the study.
* Patients scheduled for minor surgery.
* Patients with an ASA score 1 or 5.
* Patients due for outpatient surgery.
* Patients due for surgery under local or locoregional anesthesia.
* Impossibility of 28-day follow-up.
* Patients participating in interventional research involving human subjects.
* Patients in an exclusion period determined by another study.
* Patients under court protection, guardianship or curatorship.
* Patients for whom it is impossible to provide clear information.
* Pregnant, parturient or breast-feeding patients.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1028 (Actual)
Dates: Start 2024-02-05 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of death after surgery in the control group | Day 28
  YES/NO
Occurrence of death after surgery in the experimental group | Day 28
  YES/NO
Occurence of acute myocardial infarction after surgery in the control group | Day 28
  YES/NO
Occurence of acute myocardial infarction after surgery in the experimental group | Day 28
  YES/NO
Occurence of arterial or venous thrombosis after surgery in the control group | Day 28
  YES/NO
Occurence of arterial or venous thrombosis after surgery in the experimental group | Day 28
  YES/NO
Occurence of a stroke after surgery in the control group | Day 28
  YES/NO
Occurence of a stroke after surgery in the experimental group | Day 28
  YES/NO
Postoperative cardiogenic shock (requiring diuretic, epinephrine or dobutamine infusion) in the control group | Day 28
  YES/NO
Postoperative cardiogenic shock (requiring diuretic, epinephrine or dobutamine infusion) in the experimental group | Day 28
  YES/NO
Severe acute hypotension (defined as mean arterial pressure < 50 mmHg) in the control group | Day 28
  YES/NO
Severe acute hypotension (defined as mean arterial pressure < 50 mmHg) in the experimental group | Day 28
  YES/NO
Cardiac arrhythmia (de novo atrial fibrillation, atrial flutter, ventricular tachycardia, ventricular fibrillation) in the control group | Day 28
  YES/NO
Cardiac arrhythmia (de novo atrial fibrillation, atrial flutter, ventricular tachycardia, ventricular fibrillation) in the experimental group | Day 28
  YES/NO
Postoperative episodes of sepsis and infections (according to the 2001 international definitions of sepsis) in the control group | Day 28
  YES/NO
Post-operative respiratory complications: defined as the need for intubation and/or non-invasive ventilation in the event of respiratory failure in the control group | Day 28
  YES/NO
Acute kidney injury in the control group: KDIGO criteria and renal replacement therapy. Baseline serum creatinine is obtained from the preoperative blood sample; | Day 28
  YES/NO
Acute kidney injury in the experimental group: KDIGO criteria and renal replacement therapy. Baseline serum creatinine is obtained from the preoperative blood sample; | Day 28
  YES/NO
Surgical complications in the control group: need for re-operation for any reason and radiological intervention for abscess drainage | Day 28
  YES/NO
Surgical complications in the experimental group: need for re-operation for any reason and radiological intervention for abscess drainage | Day 28
  YES/NO
Unplanned admission or readmission to the intensive care unit: control group | Day 28
  YES/NO
Unplanned admission or readmission to the intensive care unit: experimental group | Day 28
  YES/NO

SECONDARY OUTCOMES:
Length of hospital stay : Control group | Day 28
  The length of stay in conventional hospitalization and in continuing care will be collected from the patient's record.
Length of hospital stay : Experimental group | Day 28
  The length of stay in conventional hospitalization and in continuing care will be collected from the patient's record.
Length of stay (hours) in the post-procedure care department : Control group | Day 28
  The length of stay in the post-procedure care department = discharge time - time of entry into the post-procedure care department will be recorded in hours.
Length of stay (hours) in the post-procedure care department : Experimental group | Day 28
  The length of stay in the post-procedure care department = discharge time - time of entry into the post-procedure care department will be recorded in hours.
Length of time in compliance with mean arterial pressure (MAP < 60 mm Hg) : Control group | Day 28
  The length of time in compliance with mean arterial pressure (MAP < 60 mm Hg) measured during the intervention will be recorded on the intervention report.
Length of time in compliance with mean arterial pressure (MAP < 60 mm Hg) : Experimental group | Day 28
  The length of time in compliance with mean arterial pressure (MAP < 60 mm Hg) measured during the intervention will be recorded on the intervention report.
Number of episodes of nausea/vomiting up to 12 hours after surgery: Control group | 12 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 12 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 12 hours post-operative.
Number of episodes of nausea/vomiting up to 24 hours after surgery: Control group | 24 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 24 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 24 hours post-operative.
Number of episodes of nausea/vomiting up to 48 hours after surgery: Control group | 48 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 48 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 48 hours post-operative.
Number of episodes of nausea/vomiting up to 12 hours after surgery: Experimental group | 12 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 12 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 12 hours post-operative.
Number of episodes of nausea/vomiting up to 24 hours after surgery: Experimental group | 24 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 24 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 24 hours post-operative.
Number of episodes of nausea/vomiting up to 48 hours after surgery: Experimental group | 48 hours post-surgery
  The cumulative number of episodes of nausea/vomiting up to 48 hours after surgery will be recorded based on the need to resort to an intravenous or oral anti-emetic up to 48 hours post-operative.
Post-surgical pain at 6 hours as measured by the Control group | At 6 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 6 hours as measured by the Experimental group | At 6 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 12 hours as measured by the Control group | At 12 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 12 hours as measured by the Experimental group | At 12 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 18 hours as measured by the Control group | At 18 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 18 hours as measured by the Experimental group | At 18 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 24 hours as measured by the Control group | At 24 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 24 hours as measured by the Experimental group | At 24 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 30 hours as measured by the Control group | At 30 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 30 hours as measured by the Experimental group | At 30 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 36 hours as measured by the Control group | At 36 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 36 hours as measured by the Experimental group | At 36 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 42 hours as measured by the Control group | At 42 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 42 hours as measured by the Experimental group | At 42 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 48 hours as measured by the Control group | At 48 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Post-surgical pain at 48 hours as measured by the Experimental group | At 48 hours post-surgery
  Pain intensity at rest and on mobilization will be measured on a visual analog scale (in which 0 = no pain and 10 = highest imaginable pain) every 6 hours, for up to 48 hours after surgery.
Confusion : Control group | Postoperative Day 1
  The number of episodes of confusion according to the Confusion Assessment Method, criterion 4 (disorientation) will be recorded.
Confusion : Control group | Postoperative Day 2
  The number of episodes of confusion according to the Confusion Assessment Method, criterion 4 (disorientation) will be recorded.
Confusion : Experimental group | Postoperative Day 1
  The number of episodes of confusion according to the Confusion Assessment Method, criterion 4 (disorientation) will be recorded.
Confusion : Experimental group | Postoperative Day 2
  The number of episodes of confusion according to the Confusion Assessment Method, criterion 4 (disorientation) will be recorded.
Surgical plethysmographic index : time within the defined thresholds: Control group | Day 0 immediately after surgery
  The time during which the surgical plethysmographic index is within the defined thresholds (intraoperatively after anesthetic induction): will be collected at the end of surgery (SPI between 20 and 50)
Surgical plethysmographic index : Time within the defined thresholds: Experimental group | Day 0 immediately after surgery
  The time during which the surgical plethysmographic index is within the defined thresholds (intraoperatively after anesthetic induction): will be collected at the end of surgery (SPI between 20 and 50)
Train-of-four: Time within the defined thresholds: Control group | Day 0 immediately after surgery
  The time during which the train-of-four parameters are within their defined thresholds (intraoperatively after anesthetic induction): TOF > 90% will be collected at the end of surgery
Train-of-four: Time within the defined thresholds: Experimental group | Day 0 immediately after surgery
  The time during which the train-of-four parameters are within their defined thresholds (intraoperatively after anesthetic induction): TOF > 90% will be collected at the end of surgery
State entropy: time within the defined thresholds: Control group | Day 0 immediately after surgery
  The time during which state entropy is within the defined thresholds (intraoperatively after anesthetic induction) will be collected at the end of surgery (SE between 40 and 60)
State entropy: Time within the defined thresholds: Experimental group | Day 0 immediately after surgery
  The time during which state entropy is within the defined thresholds (intraoperatively after anesthetic induction) will be collected at the end of surgery (SE between 40 and 60)
Mean arterial pressure: Time within the defined thresholds: Control group | Day 0 immediately after surgery
  The time during which the mean arterial pressure is within the defined thresholds (intraoperatively after anesthetic induction) i.e. MAP > 60 mmHg will be collected at the end of surgery
Mean arterial pressure: Time within the defined thresholds: Experimental group | Day 0 immediately after surgery
  The time during which the mean arterial pressure is within the defined thresholds (intraoperatively after anesthetic induction) i.e. MAP > 60 mmHg will be collected at the end of surgery
Monitor use in the Control group | Day 0 immediately after surgery
  Monitor use will be defined as the prevalence (in %) of patients with simultaneous placement of SE, SPI and NMT sensors for more than 90% of the total duration of general anesthesia.
Monitor use in the Experimental group | Day 0 immediately after surgery
  Monitor use will be defined as the prevalence (in %) of patients with simultaneous placement of SE, SPI and NMT sensors for more than 90% of the total duration of general anesthesia.
Compliance with intraoperative therapeutic targets in the Control group | Day 0 after surgery
  Compliance with intraoperative therapeutic targets will be defined as the prevalence (in %) of patients presenting the following triad: A SE between 40-60 more than 70% of the time of the maintenance phase of general anesthesia and an SPI between 20-50 more than 70% of the time of the maintenance phase of general anesthesia and TOF > 90% at extubation. These parameters will also be assessed individually.
Compliance with intraoperative therapeutic targets in the Experimental group | Day 0 after surgery
  Compliance with intraoperative therapeutic targets will be defined as the prevalence (in %) of patients presenting the following triad: A SE between 40-60 more than 70% of the time of the maintenance phase of general anesthesia and an SPI between 20-50 more than 70% of the time of the maintenance phase of general anesthesia and TOF > 90% at extubation. These parameters will also be assessed individually.
Participation rates: state registered anesthetic nurses | Day 28
  Participation will be defined as the presence/viewing of at least one teaching from among video (<90% video viewing) and/or anesthesia staff (paper sign-in sheet) and/or bibliography (paper sign-in sheet) and/or in situ training (paper sign-in sheet) : The overall participation rate and participation rates per learner class will be recorded.
Participation rates: anesthesiologist-resuscitation doctors | Day 28
  Participation will be defined as the presence/viewing of at least one teaching from among video (<90% video viewing) and/or anesthesia staff (paper sign-in sheet) and/or bibliography (paper sign-in sheet) and/or in situ training (paper sign-in sheet) : The overall participation rate and participation rates per learner class will be recorded.
Participation rates: interns | Day 28
  Participation will be defined as the presence/viewing of at least one teaching from among video (<90% video viewing) and/or anesthesia staff (paper sign-in sheet) and/or bibliography (paper sign-in sheet) and/or in situ training (paper sign-in sheet) : The overall participation rate and participation rates per learner class will be recorded.
Overall participation rates: state registered anesthetic nurses, anesthesiologist-resuscitation doctors and interns | Day 28
  Participation will be defined as the presence/viewing of at least one teaching from among video (<90% video viewing) and/or anesthesia staff (paper sign-in sheet) and/or bibliography (paper sign-in sheet) and/or in situ training (paper sign-in sheet) : An overall participation rate for all participants, whatever their learner class, will be recorded.
Overall satisfaction rate | Day 28
  The overall satisfaction rate will be measured on a Likert scale in which 0 = very dissatisfied and 10 = very satisfied.

OTHER OUTCOMES:
Patient's age | Day 0
  In years
Patient's weight | Day 0
  In kilos
Patient's height | Day 0
  In centimeters
Patient's body mass index | Day 0
  The patient's body mass index will be calculated according to kg/m2
Patient's ASA (American Society of Anesthesiologists) score | Day 0
  The ASA physical status classification system is a system for assessing the fitness of patients before surgery. In 1963 the American Society of Anesthesiologists adopted the five-category physical status classification system; a sixth category was later added.The score ranges from the healthiest to the least healthy patients. ASA 1 = healthy patient and ASA 6 = a patient who is declared brain dead and whose organs can be removed for donor purposes.
Patient's pre-operative comorbidities and associated treatments | Day 0
  All pre-operative comorbidities and their associated treatments will be recorded
Patient's Lee score | Day 0
  The Lee score is a prospectively validated model that predicts the risk of a cardiac event in patients undergoing noncardiac surgery. The revised cardiac risk index was developed from stable patients aged 50 years or more undergoing elective major non-cardiac procedures in a tertiary-care teaching hospital. This index can identify patients at higher risk for complications such as myocardial infarction, pulmonary edema, ventricular fibrillation or primary cardiac arrest, and complete heart block. Using a point system, patients are classified into four classes of risk in which class I patients have the lowest risk of a cardiac event and class IV have the highest risk.
Date of surgery | Day 0
  The date of surgery will be recorded
Type of surgery | Day 0
  The type of surgery will be described and recorded.
Duration of surgery | Day 0
  The duration of surgery will be recorded in minutes
Anesthesia: airway access | Day 0
  The type of airway access (intubation or laryngeal mask) will be recorded
Blood loss | Day 0
  Blood loss will be recorded in mL
Anesthesic agents | Day 0
  The type and dose of anesthesic agent used will be recorded
pre- and intraoperative haemodynamic parameters: MAP | Day 0
  Mean arterial pressure will be recorded in mmHg
pre- and intraoperative haemodynamic parameters: heart rate | Day 0
  Heart rate will be recorded in beats per minute
Patient's post-operative pain | Day 0
  The pain score (Visual Analog Scale < 3/10) and morphine pain titration will be recorded in the intensive care unit
Thromboprophylaxis | Day 0
  The treatment will be described and recorded
Antibioprophylaxis | Day 0
  The treatment will be described and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Yann GRICOURT, Doctor, Principal Investigator — Nîmes University Hospital, France; Mikael PERIN, Doctor, Principal Investigator — Nîmes University Hospital, France; Christophe BOISSON, Doctor, Principal Investigator — Nîmes University Hospital, France; Arianne Lannelongue, Doctor, Principal Investigator — Nîmes University Hospital, France
Locations (1):
- CHU de NIMES, Nîmes, France

REFERENCES:
- [Background] Gricourt Y, Bibollet G, Perin M, Vialatte PB, Forget P, Alexander B, Chasseigne V, Lefrant JY, Mezzarobba M, Cuvillon P. Exploring sevoflurane consumption and CO2 emissions of individual patients undergoing noncardiac surgery using a target-controlled sevoflurane administration system. J Clin Monit Comput. 2025 Oct 21. doi: 10.1007/s10877-025-01370-3. Online ahead of print. PMID 41118122
- [Result] Bernat M, Cuvillon P, Brieussel T, Roche M, Remacle A, Leone M, Lukaszewicz AC, Bouvet L, Zieleskiewicz L. The carbon footprint of general anaesthesia in adult patients: a multicentre observational comparison of intravenous and inhalation anaesthetic strategies in 35,242 procedures. Br J Anaesth. 2025 Jun;134(6):1620-1627. doi: 10.1016/j.bja.2025.01.043. Epub 2025 Apr 4. PMID 40187906